CLINICAL TRIAL: NCT06866743
Title: Seasonal Changes in Kidney Function Among Female Adults Post-Menopause
Brief Title: How Seasons Affect Kidney Health in Post-Menopausal Females
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Joseph Watso, Assistant Professor, Florida State University
Other Study IDs: STUDY00005199
Record Dates: First submitted 2025-02-14; First posted 2025-03-10 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Postmenopausal; Female
Keywords: Kidney Health; Post-Menopause; Heat Stress; Hydration; Older Adults; Aging; Postmenopausal Women
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Winter: Assessment of the cohort in winter 2025 (visit 1).
  Interventions: Other: There will be no intervention.
- Summer: Assessment of the cohort in summer 2025 (visit 2).
  Interventions: Other: There will be no intervention.

INTERVENTIONS:
Other: There will be no intervention. — This research focuses on examining seasonal variations in kidney function among postmenopausal females. As an observational study, our approach is non-interventional.

SUMMARY:
The investigators are assessing how seasonal changes affect kidney function biomarkers in post-menopausal women, an understudied group. While heat stress can reduce kidney function, previous research has not accounted for physical activity, diet, hydration, or sun exposure.

DETAILED DESCRIPTION:
Intense heat stress on the body can reduce kidney function. A recent study reported that blood markers of kidney function are lower among people in hotter climates. However, these data did not consider physical activity, food intake, fluid intake, time spent outdoors, or exposure to sunlight. Therefore, the investigators invite participants to help determine whether there are seasonal changes in kidney function biomarkers. This will also help the investigators understand if physical activity, food intake, fluid intake, time spent outdoors, or exposure to sunlight affect kidney function biomarkers between seasons. The investigators are studying female adults post-menopause since they are an understudied group.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥55 years old
* Self Reported as at least one year post-menopause
* Live in Tallahassee, Florida, or the surrounding area

Exclusion Criteria:

* Have a BMI of ≥30 kg/m2
* Systolic blood pressure of ≥140 and/or diastolic blood pressure ≥90 mmHg
* Self Reported Current or recent (regular use within the past six months) use of a diuretic medication
* Self Reported: Uncontrolled cardiovascular, respiratory, neurological, renal, liver, or metabolic health condition
* Current or recent (regular use within the past six months) use of tobacco, nicotine, nonsteroidal anti-inflammatory products
* No regular (≥once per week) purposeful heat exposure (e.g., sauna, spa, etc.)

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the greater Tallahassee, Florida area.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Plasma neutrophil gelatinase-associated lipocalin (NGAL) | Visit 1 (0 months) and Visit 2 (7 months)
  Changes in NGAL will be measured in blood samples using enzyme-linked immunosorbent assay.
Urinary neutrophil gelatinase-associated lipocalin (NGAL) | Visit 1 (0 months) and Visit 2 (7 months)
  Changes in NGAL will be measured in urine samples using radioimmunoassay.
Insulin-like growth factor-binding protein 7 (IGFBP7)*Tissue inhibitor of metalloproteinase-2 (TIMP-2) | Visit 1 (0 months) and Visit 2 (7 months)
  The product of Insulin-like growth factor-binding protein 7 (IGFBP7) and tissue inhibitor of metalloproteinase-2 (TIMP-2) will be measured in blood samples using enzyme-linked immunosorbent assays.

SECONDARY OUTCOMES:
estimated glomerular filtration rate (eGFR) | Visit 1 (0 months) and Visit 2 (7 months)
  eGFR will be calculated from creatinine using CKD-EPI equation.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Watso, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate data and/or material transfer agreement approvals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after completion of the trial, indefinitely
Access Criteria: A formal plan identifying the intended use of the data and proper completion of appropriate data and/or material transfer agreement approvals with the study PI and their institution.